CLINICAL TRIAL: NCT03185390
Title: Periampullary Lesions Via ERCP in Assuit University Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, emad mamdouh, Principle invvestigat, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17100192
Record Dates: First submitted 2017-06-03; First posted 2017-06-14 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: ERCP
Keywords: periampullary lesions

STUDY DESIGN:
Intervention Model Description: All cases admitted in Assuit university hospital with periampullary lesions detected by ERCP with ERCP guided biopsy or brush cytology within the period of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ERCP guided biopsy or brush cytology (Other): ERCP guided biopsy or brush cytology
  Interventions: Procedure: ERCP guided biopsy or brush cytology

INTERVENTIONS:
Procedure: ERCP guided biopsy or brush cytology — ERCP guided biopsy or brush cytology

SUMMARY:
A periampullary lesion may be begin as duodenal adenoma, ampullary adenoma, gall stone pregnant ampulla, Stricture, or periampullary lipoma, or malignant as pancreatic ductal adenocarcinoma, distal CBD cholangiocarcinoma, ampullary carcinoma and periampullary duodenal adenocarcinoma, pancreatic carcinoma.

The aim of the study is to detect incidence of different types of periampullary lesions detected by ERCP in Assuit University Hospital and the role of ERCP in early detection, diagnosis and management and diagnostic accuracy and sensitivity of biopsy and brush cytology taken by ERCP in a period of 1 years starting from June 2017 to June 2018.

DETAILED DESCRIPTION:
Periampullary lesion is defined as lesion located in 2CM around the ampulla of Vater. Periampullary lesions, identified during endoscopic retrograde cholangiopancreatography (ERCP), duodenoscopy or endoscopic ultrasonography (EUS) often present a diagnostic dilemma. Although some of these lesions represent a benign lesion, they also occur in case of malignancy. Therefore, management of periampullary lesions widely varies from observation for low-grade dysplasia to pancreaticoduodenectomy in case of invasive carcinoma. Unfortunately, endoscopic biopsies are by definition superficial and, therefore, the risk of a sample errors exists. On the other hand the similarity in presentation and the difficulty in accurate location of the origin of these lesions often leads to a diagnostic challenge. ERCP in addition to its diagnostic value it allows therapeutic procedures, such as sphincterotomy, stenting, and nasobiliary drainage. It permits sampling of pancreatic juice, bile, and brush or grasp biopsy, but endoscopic biopsies are by definition superficial and, therefore, the risk of a sample errors exists .

ERCP is an invasive procedure that requires an expert endoscopist/radiologist and a cooperative patient.

Very small tumors (< 1 cm) can be missed. A periampullary lesion may be begin as duodenal adenoma, ampullary adenoma, gall stone pregnant ampulla, Stricture, or periampullary lipoma, or malignant as pancreatic ductal adenocarcinoma, distal CBD cholangiocarcinoma, ampullary carcinoma and periampullary duodenal adenocarcinoma, pancreatic carcinoma.

The aim of the study is to detect incidence of different types of periampullary lesions detected by ERCP in Assuit University Hospital and the role of ERCP in early detection, diagnosis and management and diagnostic accuracy and sensitivity of biopsy and brush cytology taken by ERCP in a period of 1 years starting from June 2017 to June 2018.

ELIGIBILITY:
Inclusion Criteria:

* All cases admitted in Assuit university hospital with periampullary lesions detected by ERCP within the period of the study.

Exclusion Criteria:

* Cases diagnosed to have periampullary lesion and managed without ERCP

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
percentage of different types of periampullary massesand efficacy of ERCP guided biopsy calculating the number of cases correctly diagnosed by ERCP or guided biopsy | one year

SECONDARY OUTCOMES:
number of cases addmited in Assiut University Hospital with differrent types of periampullary mass diagnosed correctly by the help of ERCP | one year

CONTACTS AND LOCATIONS:
Overall Officials: morsy m morsy, professor, Study Director — prof
Locations (1):
- Assiut Univesity Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided